CLINICAL TRIAL: NCT02244099
Title: Controlled Substance Treatment Agreements in an Internal Medicine Residents' Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jared Moore, Assistant Professor - Clinical, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014H0102
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Anxiety; Chronic Pain; Opioid Use, Unspecified
Keywords: Controlled substance prescribing; Controlled substance treatment agreements; Opioid use
MeSH Terms: conditions — Anxiety Disorders; Chronic Pain | interventions — Controlled Substances

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Controlled Substance (Experimental): Consenting physicians who care for patients who have been prescribed a controlled substance, carisoprodol, or tramadol at least 3 times in the last 6 months in Martha Morehouse General Internal Medicine Resident Continuity Clinic.
  Interventions: Other: Controlled Substance

INTERVENTIONS:
Other: Controlled Substance — Patients will be identified using the reporting workbench in the EMR if they have been prescribed a controlled substance, carisoprodol, or tramadol at least 3 times in the last 6 months by one of the consenting resident physicians from Martha Morehouse General Internal Medicine Resident Continuity Clinic. Once identified, a comprehensive chart review for other important parameters based on best practice recommendations as described in the research protocol will be conducted in order to characterize the patient population for which the recommendations are being made to the physicians. Improvement in controlled substance, carisoprodol, and tramadol prescribing and adherence to the CSTA by the resident physicians will be tracked using a pre/post intervention comparison.

SUMMARY:
The purpose of this study is to characterize and improve controlled substance, carisoprodol and tramadol use in an internal medicine residents' clinic. Specific objectives of this study include:

* To measure the adherence to a controlled substance treatment agreement (CSTA) before and after implementation of a population management intervention
* To determine the number of patients on a CSTA with a discrepancy identified on a urine drug screen or an Ohio Automated Rx Reporting System (OARRS) report
* To track the number of patients on a morphine equivalent dose (MED) of ≥ 80 mg/day before and after implementation of a review intervention
* To characterize the healthcare utilization of patients taking controlled substances, carisoprodol, or tramadol by tracking the mean number of ED visits, hospital admissions, telephone calls, and clinic office visits during a 6 month period

DETAILED DESCRIPTION:
Reporting workbench will be used to generate a report from the EMR of all patients of consenting physicians prescribed a controlled substance, carisoprodol, or tramadol at least 3 times in the past 6 months. This report will also include demographics, number of ED visits in the last 6 months, hospital admissions in the last 6 months, the number of telephone calls documented in the last 6 months, the number of clinic visits in the last 6 months, the number of missed clinic visits in the last 6 months, controlled substance prescribed, directions for use, number of tabs of medication prescribed, number of refills given, order date and date of completion of urine drug screen if in last 6 months, if chronic pain is listed as a medical problem, and if controlled substance treatment agreement has been signed and scanned into EMR. For each patient of the consenting physicians, the EMR will be reviewed to track next clinic visit date, urine toxicology screen results, and if there is documentation of an Ohio Automated Rx Reporting System (OARRS) review. The MED for each patient will be obtained from the OARRS report and included on the data collection form. For any patients taking opioid substances at MED ≥ 80 mg/day a review of the appropriateness of this medication and dose based on EMR documentation will be conducted by clinic physicians and/or pharmacists. This will all be done in order to make recommendations to the resident physician based on our best practice recommended controlled substance agreement.

For all patients of the consenting physicians who have an upcoming office visit scheduled, any recommendations for improved adherence to the CSTA or change in controlled substance, carisoprodol, or tramadol prescribing based on EMR review findings will be given to the patient's physician prior to the office visit. Because this intervention is a quality improvement intervention and studies physician decision making but no direct interaction with the patient, the patient will not know this study is occurring. An EMR review after the patient's visit will be completed to track the acceptance of these recommendations leading to changes in the parameters listed in the data analysis section. Additionally, a second report will be generated from the reporting workbence 6 months after implementation of this workflow which includes all patients of the consenting physicians prescribed controlled substances, tramadol, and carisoprodol (including those on the initial report and those who are now new patients controlled substances since the time the report was generated) to characterize the improvement in these parameters for patients in clinic as a whole to track the improvement in adherence to a controlled substance treatment agreement. See study procedures in Figure 1. Data Collection will start on 8/1/14 and continue until 12/31/15.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Residents and attending physicians who work in the resident continuity practice

Exclusion Criteria:

* Age < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients Adhering to Controlled Substance Agreement | 18 months
  To measure the adherence to a controlled substance treatment agreement (CSTA) before and after implementation of a population management intervention

SECONDARY OUTCOMES:
Discrepancy on urine drug screen | 18 months
  To determine the number of patients on a CSTA with a discrepancy identified on a urine drug screen or an Ohio Automated Rx Reporting System (OARRS) report
Morphine Equivalent Review | 18 months
  To track the number of patients on a morphine equivalent dose (MED) of ≥ 80 mg/day before and after implementation of a review intervention
Healthcare Utilization | 18 months
  To characterize the healthcare utilization of patients taking controlled substances, carisoprodol, or tramadol by tracking the mean number of ED visits, hospital admissions, telephone calls, and clinic office visits during a 6 month period

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Barnes, PharmD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States